CLINICAL TRIAL: NCT05619705
Title: Effectiveness of Health Coaching to Reduce Cardiometabolic Risk in Early Home Visiting Services
Brief Title: Healthy for Two-Home Visiting (H42-HV): Health Coaching for Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00307430; 1P50MD017348-01 (NIH)
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Postpartum Weight Retention; Pregnancy Weight Gain; Overweight and Obesity; Behavior, Health
Keywords: Behavioral Intervention; Early Childhood Home Visiting; Overweight; Obesity; Postpartum; Pregnancy
MeSH Terms: conditions — Gestational Weight Gain; Overweight; Obesity; Health Behavior | interventions — Pregnancy; Postpartum Period

STUDY DESIGN:
Intervention Model Description: The design of the study is a randomized, two parallel-arm clinical trial. The investigators will be applying principles of a hybrid type 1 effectiveness-implementation randomized control trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy for Two-Health Coaching (H42) (Experimental): Those assigned to the intervention group will receive the 8 to 11 month H42 health coaching intervention in addition to usual home visiting and usual prenatal and postpartum care clinical services. Intervention duration will depend on the participant's gestational age at the of enrollment. Participants can be enrolled as early in pregnancy as 20 weeks gestation and as late as 33 weeks gestation. All participants would be enrolled for 6 months postpartum. Therefore, the minimum time in the intervention would be 8 months and maximum would be 11 months.
  Interventions: Behavioral: Healthy for Two-Health Coaching (H42)
- Maintain Health in Pregnancy and Postpartum (mHIPP) (Active Comparator): Those assigned to the "usual home visiting plus" comparison group, called maintain health in pregnancy and postpartum (mHIPP), will receive the typical, evidence-based experience in participants' home visiting program in addition to the participants' usual prenatal and postpartum care clinical services. In addition, the investigators will provide a brief (less than 5 minutes) maternal warning signs educational video that is available in English or Spanish. The video was developed for a home visiting client audience and is publicly available, https://mdmom.org/warningsigns.
  Interventions: Behavioral: Maintain Healthy in Pregnancy and Postpartum(mHIPP)

INTERVENTIONS:
Behavioral: Healthy for Two-Health Coaching (H42) — The H42-HV intervention includes health coaching calls, H42 web based app, mobile phone-based tracking.
  Arms: Healthy for Two-Health Coaching (H42)
Behavioral: Maintain Healthy in Pregnancy and Postpartum(mHIPP) — A brief video on maternal warning signs that is available in English or Spanish.
  Other Names: "Usual Home Visiting Plus"
  Arms: Maintain Health in Pregnancy and Postpartum (mHIPP)

SUMMARY:
The purpose of this study is to compare the effectiveness of H42-HV integrated into home visiting compared with usual home visiting services in reducing postpartum weight retention (difference between pre-pregnancy weight and weight at 6 months postpartum) among pregnant and postpartum participants. The overall goal is to improve long-term cardiometabolic health.

DETAILED DESCRIPTION:
There are four components of the H42-HV intervention: 1) Health coaching calls; 2) H42 web-based app for learning activities and goal setting functions; 3) Tracking of health behaviors (diet, exercise), and 4) Self-weighing (weekly). The overarching behavioral goals of the intervention are for participants to have lower postpartum weight retention at 6 months after delivery. Weight and behavioral goals will be promoted through the COACH Plan, a behavioral model guiding coaching calls, behavioral tracking targets and learning activities. Coaches will refer to home visitors for additional support and community resources, based on an established protocol.

* Telephone health coaching calls by trained health coaches. Calls start at enrollment, between 20-33-weeks gestation through 6 months postpartum. Although coaching calls will occur by phone or Zoom (~20 mins), when possible, some coach contact could occur at the time of home visits in person.
* Online interactive learning activities. Literacy adaptation ensured Learning Activities are at <5th grade reading level. All activities are translated into Spanish and culturally adapted to create a parallel program. Online learning activities contain embedded images (people and settings) that reflect the diversity of the investigators' target population, examples of activities that are readily available in the community and maximize the use of white space, large text and simple graphics to enhance readability and accessibility of the educational content. The investigators enhanced the platform to enable an interactive goal-setting functionality for participants to set health goals paced with participants' Learning Activities and calls. The online program is maintained and monitored by the study's health coach managers.
* Health behavior tracking (diet and exercise). Participants will receive specific skill-building on how to track diet and exercise behaviors via mainstream mobile app or paper/pencil, using procedures from the investigators' current trial. Coaches will be able to discuss tracking data with participants. Mainstream tracking apps are available in both Spanish and English.
* Weekly self-weighing. Participants will be asked to weigh themselves weekly at home using the participants' study scale.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, ≤33 weeks gestation
* Singleton pregnancy
* Pre pregnancy BMI≥25.0 Kg/m^2 (calculated based on self-reported pre pregnancy height and weight)
* Able to provide informed consent
* English or Spanish speaking
* Completion of screening and baseline data collection
* Willing to participate in the intervention and data collection procedure (e.g., home weights)

Exclusion Criteria:

* Type 1 diabetes or taking insulin prior to delivery
* Pregnant with multiple fetuses
* Unable to walk 1 block without pain or shortness of breath
* Not cleared by the study's clinicians or home visiting program staff
* Planning to relocate from area during next 1 year
* Active substance abuse disorder (except marijuana)
* Psychiatric or substance use related hospitalization in past 1 year
* Active eating disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in postpartum weight (retention) | Baseline and 6 months postpartum
  Difference between pre-pregnancy weight and weight at 6 months postpartum. Pre-pregnancy weight (baseline) will be self-reported and then confirmed by prenatal clinic medical records. 6 month postpartum weight will be obtained via BodyTrace study scales provided to all participants.

SECONDARY OUTCOMES:
Change in gestational weight (gain) | Baseline and immediately before delivery
  Difference between pre-pregnancy weight and delivery weight. Pre-pregnancy weight will be self-reported and then confirmed by prenatal clinic records. Delivery weight will be obtained via BodyTrace study scales provided to each participant.
Change in maternal diet as assessed by the Dietary Screener Questionnaire (DSQ) | Baseline, 37 weeks gestation, 2 months postpartum, 4 months postpartum, 6 months postpartum
  Dietary intake will be assessed using the NHANES 2009-10 Dietary Screener Questionnaire (DSQ) Eating Habits Questionnaire (28-items). Scoring equations exist to estimate daily intake of fruits/vegetables, dairy, added sugars, whole grains, and calcium.
Change in maternal physical activity as assessed by the International Physical Activity Questionnaire (IPAQ) | Baseline, 37 weeks gestation, 2 months postpartum, 4 months postpartum, 6 months postpartum
  The Short Form International Physical Activity Questionnaire contains 9 items to collect data on health-related physical activity in the past seven days. Physical activity is categorized as high (at least one hour of moderate intensity exercise daily), moderate (approximately 30 minutes of moderate intensity exercise most days), or low (not meeting the criteria of high or moderate exercise).
Maternal smoking habits as assessed by the Center for Disease Control and Prevention Pregnancy Risk Assessment Monitoring System (CDC PRAMS) | Baseline
  A four-item portion of the PRAMS survey will be utilized to determine cigarette use before and during pregnancy.
Change in breastfeeding Practice as assessed by the Center for Disease Control and Prevention Infant Feeding Practices Survey (CDC IFPS) | 2 months postpartum, 4 months postpartum, 6 months postpartum
  A 4-item portion of the CDC IFPS will be used at 2,4, and 6 months postpartum to assess current breastfeeding practice.
Breastfeeding Intention as assessed by the Center for Disease Control and Prevention Infant Feeding Practices Survey (CDC IFPS) | 37 weeks gestation
  A two-item portion of the CDC IFPS will be used to assess breastfeeding intention.
Change in maternal depression as assessed by the Edinburgh Postpartum Depression scale | Baseline, 37 weeks gestation, 2 months postpartum, 4 months postpartum, 6 months postpartum
  The Edinburgh Postpartum Depression scale is a 10-item measure assessing changes in mood over the past seven days. The last question related to suicidal ideation has been removed. Mothers who score above 13 are likely to be suffering from a depressive illness of varying severity.
Change in maternal sleep habits as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, 2 months postpartum, 4 months postpartum, 6 months postpartum
  The PSQI is a 19-item questionnaire assessing sleep habits in the past seven days. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score (0-21) and higher scores indicate worse sleep quality.
Change in maternal social support as assessed by the Functional Social Support Questionnaire (FSSQ) | Baseline, 36-38 weeks prenatal, 2 months postpartum, 4 months postpartum, 6 months postpartum
  The FSSQ is an 8-item measure that evaluates confidant support and affective support. Responses are scored 1-5 and an average is calculated based on the response from all eight items. A higher score indicates greater perceived social support.
Maternal healthcare utilization as assessed by Medicaid data extraction | Up to 6 months after delivery
  Postpartum OBGYN visit and primary care provider visit by six months.
Infant healthcare utilization as assessed by Medicaid data extraction | Up to 6 months after delivery
  Well-child visit appointments through six months of life.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Bower, PhD, MSN/MPH, Principal Investigator — Johns Hopkins School of Nursing; Wendy Bennett, MD,MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin LM, McKinney CD, Escobar Acosta L, Coughlin JW, Jeffers NK, Solano-Umana A, Carson KA, Wang NY, Bennett WL, Bower KM. Remote Lifestyle Intervention to Reduce Postpartum Weight Retention: Protocol for a Community-Engaged Hybrid Type I Effectiveness-Implementation Randomized Controlled Trial. JMIR Res Protoc. 2025 Jan 7;14:e62847. doi: 10.2196/62847. PMID 39773922